CLINICAL TRIAL: NCT01249651
Title: An 8-week, Open Label, Multicentre Study to Assess the Efficacy of Esomeprazole 40 mg Once Daily in Subjects With Continuing Symptoms of Heartburn Following Treatment With a Previous Rabeprazole.
Brief Title: To Assess the Efficacy of Esomeprazole 40 mg Once Daily in Subjects Who Still Had Heartburn After Receiving Rabeprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D961HL00001
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-06

CONDITIONS: Heartburn
Keywords: Patients, Single
MeSH Terms: conditions — Heartburn | interventions — Esomeprazole

ARMS (1):
- 1 (Other): One arm: esomeprazole 40 mg
  Interventions: Drug: esomeprazole 40 mg

INTERVENTIONS:
Drug: esomeprazole 40 mg — esomeprazole 40 mg once daily, 8 weeks
  Other Names: No comparator

SUMMARY:
Administration of esomeprazole 40 mg to subjects who still had heartburn after receiving rabeprazole 20 mg once daily for 4 to 8 weeks will result in statistically significant improvement of heartburn after 8-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20 years or more
* Documented history of reflux esophagitis verified by endoscopy in the past, including the grade of Los Angeles (LA) classification (Lundell LR et al 1999) before treatment
* Ongoing (until date of Visit 1) treatment with rabeprazole 20 mg, given once daily, for a period of 4 to 8 weeks. The subject must take Rabeprazole at least 4 days a week in the past 7 days prior to Visit 1.
* Persisting symptoms of heartburn during the past 7 days prior to Visit 1, judged by the investigator(s) as follows: At least 2 days with moderate (i.e. discomfort sufficient to cause interference with normal activities) to severe symptoms (i.e. incapacitating, with inability to perform normal activities) OR At least 4 days with symptoms including mild ones (i.e. awareness of sign or symptom, but easily tolerated).
* The subject needs to be able to understand and read the official languages of the country.

Exclusion Criteria:

* Use of other PPIs and/or H2RA during rabeprazole treatment
* Previous use of esomeprazole 40 mg during the 12 weeks before enrolment
* Current or historical evidence of gastrointestinal pathology
* History, signs or symptoms of clinically significant or uncontrolled cardiovascular, pulmonary, renal, endocrine, hematologic, neurologic, psychiatric pancreatic or hepatic disease as judged by the investigator to interfere with the conduct of the study, the interpretation of study results, subject compliance, or the health of the subject during the study.
* Documented upper gastrointestinal surgery such as gastric resection, vagotomy and/or pyloroplasty, hiatus hernia surgery or fundoplication. Note: endoscopic polypectomy, endoscopic mucosal resection, endoscopic submucosal dissection or simple suturing of an ulcer are not exclusion criteria.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Date, MD, PhD, Study Director — AstraZeneca KK Corporate Communications
Locations (1):
- Research Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled on 23 November 2010. Last participant completed on 11 June 2011. Out of 101 enrolled participants, 100 participants (target was 100) received esomeprazole 40 mg. All of the participants were included in safety analysis set and 96 out of the 100 participants were included in the full analysis set for efficacy analyses.
Pre-assignment Details: Participants with a history of reflux oesophagitis and with continuing heartburn after previous treatment with rabeprazole 20 mg were included in this study.
Period: Overall Study
Arm/Group | Esomeprazole 40 mg
Started | 101 (Enrolled)
Completed | 94 (Completed the 8-week treatment period)
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Sponsor Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esomeprazole 40 mg
Number analyzed (Participants) | 101
Age Continuous [Mean (Standard Deviation); unit: Year] | 51.2 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in the Frequency of Heartburn During the 7-day Period Prior to the 8 Week Visit (Visit 3) Compared to the Frequency of Heartburn During the 7-day Period Prior to Baseline (Visit 1)
Description: The number of days with heartburn during the 7-day period prior to the 8 week visit (Visit 3) was compared to the number of days with heartburn during the 7-day period prior to baseline (Visit 1). The difference in the number of days with heartburn from baseline to 8 weeks was analysed.
Time Frame: Baseline to 8 weeks
Population: Full analysis set (96 participants)
Measure: Mean (Standard Deviation); unit: Number of days
Groups:
- Arm 1 - Esomeprazole 40 mg: esomeprazole 40 mg once daily, 8 weeks
Arm/Group | Arm 1 - Esomeprazole 40 mg
Number analyzed (Participants) | 96
Number of days | -3.3 (2.36)
Statistical Analysis 1: Comparison: Arm 1 - Esomeprazole 40 mg; Wilcoxon signed-rank test was used to check whether the change in the frequency of heartburn during the 7-day period prior to the 8 week visit (Visit 3) compared to the frequency of heartburn during the 7-day period prior to baseline (Visit 1) was statistically significant or not; Test type: Superiority or Other; p < 0.001, Wilocoxon signed-rank test

2. Secondary Outcome: Change in the Frequency of Heartburn During the 7-day Period Prior to the 4 Week Visit (Visit 2) Compared to the Frequency of Heartburn During the 7-day Period Prior to Baseline (Visit 1)
Description: The number of days with heartburn during the 7-day period prior to the 4 week visit (Visit 3) was compared to the number of days with heartburn during the 7-day period prior to baseline (Visit 1). The difference in the number of days with heartburn from baseline to 4 weeks was analysed.
Time Frame: Baseline and 4 weeks
Population: 92 Participants in the Full analysis set (96 participants) had data of heartburn.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Arm 1 - Esomeprazole 40 mg
Number analyzed (Participants) | 92
Number of days | -2.6 (2.82)

3. Secondary Outcome: Change in the Maximum Severity of Heartburn During the 7-day Period Prior to the 4 Week Visit (Visit 2) Compared to the Frequency of Heartburn During the 7-day Period Prior to Baseline (Visit 1)
Description: Maximum severity of heartburn during 7 days at baseline and at 4 weeks was obtained (None, Mild, Moderate, Severe). If the value at 4 weeks was better than at baseline in a participant, the participant was s categorized into "Improved". If the value was same, then categorised into "Unchanged". If the value was worsened, categorised into "Worsened".
Time Frame: Baseline and 4 weeks
Population: 92 Participants in the Full analysis set (96 participants) had data of heartburn at week 4.
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Esomeprazole 40 mg
Number analyzed (Participants) | 92
Participants
  Improved | 77
  Unchanged | 14
  Worsened | 1

4. Secondary Outcome: Change in the Maximum Severity of Heartburn During the 7-day Period Prior to the 8 Week Visit (Visit 3) Compared to the Frequency of Heartburn During the 7-day Period Prior to Baseline (Visit 1)
Description: Maximum severity of heartburn during 7 days at baseline and at 8 weeks was obtained (None, Mild, Moderate, Severe). If the value at 8 weeks was better than at baseline in a participant, the participant was s categorized into "Improved". If the value was same, then categorised into "Unchanged". If the value was worsened, categorised into "Worsened".
Time Frame: Baseline to 8 weeks
Population: Full analysis set (96 participants)
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Esomeprazole 40 mg
Number analyzed (Participants) | 96
Participants
  Improved | 83
  Unchanged | 12
  Worsened | 1

ADVERSE EVENTS:
Arm/Group | Esomeprazole 40 mg
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 2/100
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 40 mg (N=100)
Nasopharyngitis (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.